CLINICAL TRIAL: NCT06539403
Title: Thinking About Memory: How Confident Are You in Your Memory, and Does it Change With Age? Investigating Memory Ability and Confidence in Those Attending Memory Clinics.
Brief Title: Thinking About Memory: How Confident Are You in Your Memory, and Does it Change With Age?
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 316787
Record Dates: First submitted 2024-04-08; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment; Subjective Cognitive Decline
Keywords: Memory; Metacognition; Mild Cognitive Impairment; Subjective Cognitive Decline; Ageing
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients Diagnosed with Mild Cognitive Impairment: Two-three hour (including breaks) behavioural testing session: taking part in memory tasks and completing questionnaires
  Interventions: Behavioral: Memory tasks
- Participants attending Memory Clinics who do not have diagnosis of Mild Cognitive Impairment: Two-three hour (including breaks) behavioural testing session: taking part in memory tasks and completing questionnaires
  Interventions: Behavioral: Memory tasks
- Healthy Control Participants: Two-three hour (including breaks) behavioural testing session: taking part in memory tasks and completing questionnaires
  Interventions: Behavioral: Memory tasks

INTERVENTIONS:
Behavioral: Memory tasks — Naturalistic Episodic Memory encoding: Participants will play short sessions of 3 board games with the researcher. The board games include Ludo, Snakes & Ladders and Solitaire. Participants will play each boardgame for around 5 min. They will wear a head camera while playing the games.
  Later participants will be tested on their memory of the naturalistic episodic memory task, a semantic memory task (memory of facts) and a perceptual task. Each task will consist of 2-3 sub-tasks of around 30 trials. These tasks will all take place on the computer and will take 30-40 minutes in total. In each trial participants will choose between two options. For example: Which of these two images is taken from your head camera? What colour piece did you use in 'snakes and ladders'?. After they choose their answer, they will report how confident they are in their choice. At the end of each task, they will be asked to report how well they think they performed on the task overall.

SUMMARY:
Memory and our own beliefs and confidence in our ability to remember are important for our daily lives. For example, low confidence may hold us back from doing certain tasks, whereas misplaced high confidence in our memories may lead us to false beliefs about what has happened in the past.

However, it is not fully understood how people form their beliefs about their memory abilities. These beliefs we hold about how good our memory is are form of evaluation of our own abilities known as 'metacognition'. The purpose of this study is to better understand how individuals, both with and without diagnosed memory difficulties, perform memory tasks and examine whether their metacognition of their memory performance depends on the type of memory task. That is, the study examines metacognition for different forms of memory; for example memory of our experienced life events as compared to memory for facts. There is still much more to learn about how individuals experience and think about their memories and memory abilities; and understanding this is important as some evidence suggests that good metacognition is associated with better outcomes after diagnosis of cognitive impairment. Understanding metacognitive beliefs about memory could be a route to earlier diagnosis and enable us to identify people who are likely to develop dementia.

DETAILED DESCRIPTION:
Our confidence in our memory ability is important for our wellbeing, especially in older age as many of us begin to fear developing dementia. The ability to judge our own cognitive abilities, such as our memory, is called metacognition. The confidence we have in our memory can be affected by changes in these metacognitive skills. Many older individuals are referred to memory clinics because they believe that their memory ability has decreased. Some individuals with these memory complaints, but without dementia, demonstrate signs of impairment to their thinking processes when tested by clinicians and are given the diagnosis Mild Cognitive Impairment (MCI). Others show no impairment when tested and are given the diagnosis Subjective Cognitive Decline (SCD). A sparse amount of research has investigated the metacognitive abilities of these groups of individuals; both those with MCI and those with SCD. Investigation of these abilities is important as some work suggests that good metacognition is associated with better symptom outcomes (Chi et al., 2022; Zhuang et al., 2022). Understanding the mechanisms underlying metacognitive beliefs about memory could be a route to earlier diagnosis and enable us to identify people who are likely to develop dementia. In this study we will recruit individuals with both MCI or SCD and age-matched controls, who do not feel that they have memory impairments, in order to investigate their metacognitive beliefs about their memory abilities.

Primary Objective: The primary objective of the study is to measure whether metacognitive judgements of memory performance differ between older healthy individuals and patients who have been referred to memory clinics. The study will include patients diagnosed with Mild Cognitive Impairment (MCI) and those with Subjective Cognitive Decline (SCD) to examine how they judge their ability to remember, compared to healthy older individuals.

To achieve this objective, the following will be assessed:

How do people rate their own memory in daily life and does this vary across different memory domains? (this is known as self-belief)

How do people rate their ability to complete the tasks we ask them to take part in? (known as global metacognition)

How confident are people in their memory when they take part in a memory task? (known as local metacognition)

Are there differences in 1), 2) and 3) between individuals with and without memory complaints?

The 'global' and 'local' metacognition examined in 2) and 3) will be compared across different types of cognitive task. The cognitive tasks assess semantic and episodic memory and visual perception. This will allow examination of the following:

Are there differences in global (how confident they think about completing the task overall) and local metacognition (hoe confident they are for each response they give) between the different tasks, e.g., between semantic memory and episodic memory?

What is the relationship between self-beliefs, global and local metacognition? Examined through a self-belief questionnaire at the start and the self-rated confidence values given throughout the tasks.

Are there differences in 5) and 6) between individuals with and without memory complaints?

Secondary objective:

Are there differences in cognitive performance between those with and without memory complaints? This is assessed through the scores people achieve on the tasks used - rather than on the confidence ratings people give while completing the tasks.

Are there differences in cognitive performance between the three types of task? Performance will be examined for each individual task separately (e.g., spatial information and object information maintenance - both of which are art of the episodic memory battery.

Does dementia worry moderate the metacognitive processes of the individuals? This will be assessed by examining responses given in the Dementia Worry questionnaire and comparing their level of dementia worry (high, medium, low) to the confidence ratings they give throughout.

ELIGIBILITY:
Inclusion Criteria:

* In age range given above
* Referred to memory clinic
* No other current psychiatric or neurological disorders, except for migraine
* Can understand verbal or written information given in English.

Exclusion Criteria:

* Outside age range given above
* If they have a diagnosis of dementia and/or inability to provide informed consent.
* Diagnosis of other neurological and/ or psychiatric problems.
* Healthy participants will be excluded if they have participated in the previous study (King's REC ref: HR/DP-21/22-302230), as this study is a continuation of that.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants will be identified through the South London and Maudsley (SLaM) NHS memory clinics, the Joint Dementia research internal database REDCap and the Brain health Clinic at King's College London. Service users who satisfy the inclusion criteria of the study will be identified by clinics and research teams in the respective services and informed about the study. If participants give consent to contact (provided by the services mentioned above), the research team will contact the participants through email and provide further information about the study. Should the participant agree to participate, they will be offered to come to the test lab at King's College London Guy's campus.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Do metacognitive judgements of memory performance differ between older healthy individuals and patients who have been referred to memory clinics? | Assessed in single 2-3 hour session per participant
  The following will be assessed:
  1. How do people rate their own memory overall? Known as self-belief. This is questionnaire in which they rate their own memory on a scale of 1-5; with 1 being 'extremely bad' and 5 being 'extremely good'.
  2. How do people rate their ability to complete the tasks? Known as global metacognition. Before and after each task they will rate how good they think they will be, or were, at the task. Also rated on the scale of 1-5.
  3. How confident are people in their memory while taking part in a memory task? Known as local metacognition. After each trial of the task, they will answer 'how confident are you that you were correct in that trial?'; again on the same scale of 1-5.
  All scales in the primary outcome measure are designed for this set of tasks. The ratings given will be pooled into a level of self-belief; global metacognition and local metacognition for each person. All of which are needed to evaluate the primary outcome measure.
Do metacognitive judgements of memory performance vary across different types of cognitive information (e.g., episodic versus semantic) individuals make their confidence judgements on? | Assessed in single 2-3 hour session per participant
  The following will be assessed:
  1. How confident are people in their memory while taking part in the memory tasks that probe the event they experienced (episodic memory)? After each trial of these tasks, they will answer 'how confident are you that you were correct in that trial?'; again on the same scale of 1-5.
  2. How confident are people in their memory while taking part in tasks of general knowledge (semantic memory)? After each trial of the task, they will answer 'how confident are you that you were correct in that trial?'; again on the same scale of 1-5.
  These tasks are the same as those referred to in Outcome 1 but this is to indicate that they will also be separately analysed.

SECONDARY OUTCOMES:
Are there differences in cognitive performance between those with and without memory complaints? | Assessed in single 2-3 hour session per participant
  The secondary outcome consists of the data for task performance itself - rather than confidence ratings described above. That is during the episodic memory tasks and semantic memory tasks they will be either correct or incorrect on each trial and so a proportion of trials correct will be calculated for each memory domain. There are up to 90 trials per domain, so proportion correct is X/90 for each domain.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We may share outcome measures with the CARE network at KCL as they are putting us in contact with their healthy control participant database.

REFERENCES:
- [Background] Chi SY, Rabin LA, Aronov A, Fogel J, Kapoor A, Wang C. Differential focal and nonfocal prospective memory accuracy in a demographically diverse group of nondemented community-dwelling older adults. J Int Neuropsychol Soc. 2014 Nov;20(10):1015-27. doi: 10.1017/S1355617714000964. Epub 2014 Nov 17. PMID 25401793
- [Background] Chi SY, Chua EF, Kieschnick DW, Rabin LA. Retrospective metamemory monitoring of semantic memory in community-dwelling older adults with subjective cognitive decline and mild cognitive impairment. Neuropsychol Rehabil. 2022 Apr;32(3):429-463. doi: 10.1080/09602011.2020.1831552. Epub 2020 Oct 26. PMID 33106082
- [Background] Jenkins A, Tree J, Tales A. Distinct Profile Differences in Subjective Cognitive Decline in the General Public Are Associated with Metacognition, Negative Affective Symptoms, Neuroticism, Stress, and Poor Quality of Life. J Alzheimers Dis. 2021;80(3):1231-1242. doi: 10.3233/JAD-200882. PMID 33646150
- [Background] Zhuang, K., Chen, X., Cassady, K. E., Baker, S. L., & Jagust, W. J. (2021). Metacognition, cortical thickness, and tauopathy in aging. bioRxiv, 2021.2010.2027.466146. https://doi.org/10.1101/2021.10.27.466146